CLINICAL TRIAL: NCT00209859
Title: Combination Treatment With Methotrexate and Cyclosporine in Early Rheumatoid Arthritis.
Brief Title: Methotrexate and Cyclosporine in Treatment of Early Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 232-002
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Cyclosporine

INTERVENTIONS:
Drug: Methotrexate
Drug: Intraarticular betamethasone
Drug: Cyclosporine/placebo-cyclosporine

SUMMARY:
To investigate whether cyclosporine, added to methotrexate and steroid, increases the possibility of inflammatory management early in the disease; furthermore to investigate the possible steroid-sparing effect of cyclosporine in patients with recently diagnosed rheumatoid arthritis.

DETAILED DESCRIPTION:
Design: Multicentre, prospective, randomised, double-blind study with parallel design.

Selection of patients: Patients with recently diagnosed rheumatoid arthritis (less than 6 months of persistent synovitis).

ELIGIBILITY:
Inclusion Criteria:

* Synovitis in at least 2 joints.
* Compliance with the ACR criteria for RA.
* Duration of no more than 6 months (from the first anamnestic non-traumatic synovitis of at least 6 weeks' duration).
* Informed consent.

Exclusion Criteria:

* Age less than 18 years or more than 75 years
* Lack of co-operability.
* Previous treatment with DMARD
* Corticosteroid treatment during the preceding 4 weeks.
* Contra indications for the treatments (awaiting the recommendations from Novartis)
* Previous or present malignant or premalignant disease
* Poorly regulated hypertension
* Impaired renal function
* Immuno defective diseases, including HIV
* Cardiac or pulmonary insufficiency
* Serious arteriosclerosis
* Serious granulocytopenia or thrombocytopenia
* Impaired liver function (liver enzymes more than twice the highest normal limit).
* Alcohol consumption of more than 3 drinks a week.
* Poorly controlled epilepsy
* Lack of contraception in fertile patients
* Pregnancy and lactation
* Psoriasis
* Poorly regulated diabetes
* Anticoagulant treatment
* Known allergy to the medicine
* Medicamental interactions
* Other inflammatory rheumatic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 1998-10; Study Completion 2007-11

PRIMARY OUTCOMES:
ACR20 response

SECONDARY OUTCOMES:
ACR remission (modified)
Cumulated dose of glucocorticoids
Development of erosions
Development of osteopenia

CONTACTS AND LOCATIONS:
Overall Officials: Merete L Hetland, MD, PhD, Principal Investigator — Hvidovre Univervsity Hospital; Kim Hørslev-Petersen, MD, DSc, Principal Investigator — Rheumatism Hospital Graasten
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Herly M, Stengaard-Pedersen K, Vestergaard P, Ostergaard M, Junker P, Hetland ML, Horslev-Petersen K, Ellingsen T. The D-vitamin metabolite 1,25(OH)2 D in serum is associated with disease activity and Anti-Citrullinated Protein Antibodies in active and treatment naive, early Rheumatoid Arthritis Patients. Scand J Immunol. 2018 Sep;88(3):e12704. doi: 10.1111/sji.12704. Epub 2018 Aug 22. PMID 30048002
- [Derived] Herly M, Stengaard-Pedersen K, Horslev-Petersen K, Hetland ML, Ostergaard M, Christensen R, Logstrup BB, Vestergaard P, Podenphant J, Junker P, Ellingsen T. Association between baseline vitamin D metabolite levels and long-term cardiovascular events in patients with rheumatoid arthritis from the CIMESTRA trial: protocol for a cohort study with patient-record evaluated outcomes. BMJ Open. 2017 Apr 8;7(4):e014816. doi: 10.1136/bmjopen-2016-014816. PMID 28391237
- [Derived] Hetland ML, Ostergaard M, Ejbjerg B, Jacobsen S, Stengaard-Pedersen K, Junker P, Lottenburger T, Hansen I, Andersen LS, Tarp U, Svendsen A, Pedersen JK, Skjodt H, Ellingsen T, Lindegaard H, Podenphant J, Horslev-Petersen K; CIMESTRA study group. Short- and long-term efficacy of intra-articular injections with betamethasone as part of a treat-to-target strategy in early rheumatoid arthritis: impact of joint area, repeated injections, MRI findings, anti-CCP, IgM-RF and CRP. Ann Rheum Dis. 2012 Jun;71(6):851-6. doi: 10.1136/annrheumdis-2011-200632. Epub 2012 Feb 1. PMID 22302316
- [Derived] Christensen AF, Horslev-Petersen K, Christgau S, Lindegaard HM, Lottenburger T, Junker K, Hetland ML, Stengaard-Pedersen K, Jacobsen S, Ellingsen T, Andersen LS, Hansen I, Skjodt H, Pedersen JK, Lauridsen UB, Svendsen AJ, Tarp U, Podenphant J, Heegaard NH, Vestergaard A, Jurik AG, Ostergaard M, Junker P. Uncoupling of collagen II metabolism in newly diagnosed, untreated rheumatoid arthritis is linked to inflammation and antibodies against cyclic citrullinated peptides. J Rheumatol. 2010 Jun;37(6):1113-20. doi: 10.3899/jrheum.091265. Epub 2010 May 1. PMID 20436079
- [Derived] Christensen AF, Sorensen GL, Horslev-Petersen K, Holmskov U, Lindegaard HM, Junker K, Hetland ML, Stengaard-Pedersen K, Jacobsen S, Lottenburger T, Ellingsen T, Andersen LS, Hansen I, Skjodt H, Pedersen JK, Lauridsen UB, Svendsen A, Tarp U, Podenphant J, Vestergaard A, Jurik AG, Ostergaard M, Junker P. Circulating surfactant protein -D is low and correlates negatively with systemic inflammation in early, untreated rheumatoid arthritis. Arthritis Res Ther. 2010;12(2):R39. doi: 10.1186/ar2948. Epub 2010 Mar 8. PMID 20211020
- [Derived] Hetland ML, Ejbjerg B, Horslev-Petersen K, Jacobsen S, Vestergaard A, Jurik AG, Stengaard-Pedersen K, Junker P, Lottenburger T, Hansen I, Andersen LS, Tarp U, Skjodt H, Pedersen JK, Majgaard O, Svendsen AJ, Ellingsen T, Lindegaard H, Christensen AF, Vallo J, Torfing T, Narvestad E, Thomsen HS, Ostergaard M; CIMESTRA study group. MRI bone oedema is the strongest predictor of subsequent radiographic progression in early rheumatoid arthritis. Results from a 2-year randomised controlled trial (CIMESTRA). Ann Rheum Dis. 2009 Mar;68(3):384-90. doi: 10.1136/ard.2008.088245. Epub 2008 Apr 3. PMID 18388160